CLINICAL TRIAL: NCT01353183
Title: Analysis of the Enteric Nervous System Using Colonic Biopsies: a Useful Biomarker for the Differential Diagnosis of Parkinsonian Syndromes?
Brief Title: Analysis of the Enteric Nervous System Using Colonic Biopsies
Acronym: ColoBioParker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/4-U; ID RCB 2010-A00632-37 (Registry Identifier: 2010-A00632-37)
Record Dates: First submitted 2011-01-31; First posted 2011-05-12 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: biopsies, enteric nervous system, biomarker
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colonic biopsies (Experimental): Colonic biopsies obtained during the course of colonoscopy or rectosigmoidoscopy
  Interventions: Procedure: colonoscopy or rectosigmoidoscopy

INTERVENTIONS:
Procedure: colonoscopy or rectosigmoidoscopy — Usual procedure

SUMMARY:
The aim of this project is to develop an original biomarker for Parkinson's disease (PD) and other parkinsonian syndromes (multiple system atrophy and progressive supranuclear palsy) based upon the detection of pathological alpha-synuclein species in routine colonoscopic biopsies.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patients aged 50-80 year old, both genders
* Parkinson's disease patients
* Multiple system atrophy patients
* Progressive supranuclear palsy patients
* Controls: patient at risk of colic cancer for whom a colonoscopy is required
* Patients who signed the informed consent

Controls

* Patients aged 50 to 80 year-old for whom a rectosigmoidoscopy or a colonoscopy is required for colorectal screening
* Patients who signed the informed consent
* Health care beneficiary

Exclusion Criteria:

Patients

* Colonic disorder (except non-complicated diverticular disease)
* Other neurological disorder than parkinsonism
* Patients treated with either platelet antiaggregants, anticoagulants or with a known coagulation disorder
* Patients with a cognitive impairment that preclude them from understanding the informed consent
* Patients placed under legal guardianship

Controls

* Neurodegenerative disorders such as Parkinson's disease, Alzheimer's disease or other dementia, amyotrophic lateral sclerosis...
* Functional bowel disorder such as irritable bowel syndrome
* Patients with a cognitive impairment that preclude them from understanding the informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Presence of alpha-synuclein aggregates in colonic biopsies using immunohistochemistry | 3 months
  Colonic biopsies are obtained during the course of colonoscopy or rectosigmoidoscopy.

SECONDARY OUTCOMES:
Presence of alpha-synuclein aggregates in colonic biopsies using 2D electrophoresis | 3 months
  Colonic biopsies are obtained during the course of colonoscopy or rectosigmoidoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: DERKINDEREN Pascal, Professor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France